CLINICAL TRIAL: NCT05989295
Title: The Efficacy, Safety and Acceptability of a Probiotic in Reducing the Scorad Index in Children With Atopic Skin
Brief Title: A Probiotic That Reduces Atopic Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Collaborators: Methodex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: WK2023002
Record Dates: First submitted 2023-07-17; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Atopic Skin; Children
Keywords: atopic skin;; eczema;; child population;; probiotic
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): 2.0 g maltodextrin /sachet； Take one sachet a day before meals. Dilute in water； Store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: probiotic LRa05
- Probiotic group (Active Comparator): (2B CFU/sachet) Lactobacillus rhamnosus LRa05 and maltodextrin Take one sachet a day before meals. Dilute in water； Store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: probiotic LRa05

INTERVENTIONS:
Dietary Supplement: probiotic LRa05 — treatment about 12 weeks

SUMMARY:
To assess the efficacy and safety of the use of probiotics as food supplements in reducing the SCORAD index in children with atopic skin compared with placebo. This is a randomized, placebo-controlled, double-blind clinical trial with 2 parallel groups, which will include 32 patients who attend some of the research centers. Patients will be randomized into one of the 2 study groups (allocation ratio 1: 1): Experimental group (Lactobacillus rhamnosus LRa05) and placebo group (placebo). The reduction of the SCORAD index, the number of sprouts in 12 weeks, the days of use of topical corticosteroids and one valuations of the skin condition (hydration).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with atopic dermatitis in the sprouts phase with a moderate SCORAD index (16-40).
2. Patients aged 2-14 years.

Exclusion Criteria:

* Patients intolerant to gluten, lactose or cow's milk protein.
* Patients who change the type of diet during the study to improve their atopic dermatitis.
* Patients with atopic dermatitis in remission phase (absence of sprouts and with SCORAD index = 0).
* Patients with an allergy or intolerance to any of the ingredients in the formulation of the product under study.
* Patients taking immunomodulators, topical or oral antibiotics, topical or oral antihistamines, oral corticosteroids or antineoplastics.
* Subjects whose condition does not make them eligible for the study, according to the investigator.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
the outbreaks of atopic skin | 12 weeks
  use the SCORAD index to measure the outbreaks of atopic skin

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - CAP Alhambra of Hospitalet de Llobregat, Barcelona
  - CAP La Mina Carrer Mar Sant Adrià de Besos, Barcelona

IPD SHARING:
Plan to Share IPD: No